CLINICAL TRIAL: NCT06237751
Title: Preoperative Sildenafil Administration for Hepatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Chenzhou (Other)
Responsible Party: Principal Investigator, zhiming zhang, chief, First People's Hospital of Chenzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023139
Record Dates: First submitted 2023-12-03; First posted 2024-02-01 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Central Venous Pressure; Hepatectomy; Hemodynamics Instability; Sildenafil
Keywords: Sildenafil Citrate; Hepatectomy; Laparoscopy; Low central venous pressure; Study protocol
MeSH Terms: interventions — Sildenafil Citrate; Nitroglycerin

STUDY DESIGN:
Intervention Model Description: The investigators planned a study to evaluate the feasibility and efficacy of sildenafil citrate by comparing 2 groups of patients, the first without the drug and the second with 25 mg of sildenafil citrate.1) Feasibility and efficacy were assessed by comparing the amount of intraoperative bleeding, the effect of CVP, and the surgeon's operative field grading.2) Liver and renal function indexes, length of hospitalization, hospitalization costs, and postoperative complications were assessed by comparing patients' preoperative, 1d postoperative, 3d postoperative, and 7d postoperative occurrence, to assess the safety of its clinical application.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- calcium tablet (Other): calcium tablet
  Interventions: Drug: Sildenafil 100 MG

INTERVENTIONS:
Drug: Sildenafil 100 MG — Sildenafil 100mg orally half an hour before surgery
  Other Names: nitroglycerine

SUMMARY:
Hepatectomy is an important treatment for liver diseases, and bleeding is one of the most common complications during dissection of the liver parenchyma. The Control Low Central Venous Pressure (CLCVP) technique is currently one of the most important techniques to control intraoperative bleeding. It mainly consists of fluid restriction, position adjustment, and the use of vasodilators. However, these measures focus on decreasing CVP by reducing the volume of return blood, and less attention is paid to factors such as pulmonary vascular resistance and cardiac function. Sildenafil, known as Viagra, is currently used to treat erectile dysfunction and pulmonary hypertension in men. Its action inhibits phosphodiesterase-5 (PDE-5) and increases cGMP levels, leading to smooth muscle relaxation and vasodilation. Its pharmacological properties provide potential value for the treatment of many diseases. However, few studies have been conducted both domestically and internationally on the use of sildenafil citrate in liver resection related to CLCVP. This study aims to investigate the influence of preoperative oral administration of Sildenafil Citrate combined with IPM on IBL and surgical results during open or laparoscopic hepatectomy, as well as its safety and feasibility. It is expected to provide an innovative management optimization plan for reducing the bleeding in hepatectomy and to provide empirical support for the potential value of Sildenafil Citrate or Sildenafil-like drugs in improving the safety and quality of perioperative hepatectomy patients.

DETAILED DESCRIPTION:
1. Feasibility/Effectiveness evaluation indicators:

   Primary outcomes：
   * Intraoperative blood loss: To quantify the IBL by calculating the amount of blood in the suction bottle (actual blood loss amount - saline irrigation amount) and the weight of the gauze blood pad ((weight of the gauze block after blood absorption in g - weight of the gauze block before blood absorption in g) / 1.054 (average density of blood in g/ml)).
   * The classification of the surgical field: At T3 and T4, the surgeon will rate and score the liver surgical field according to Table 2. If the score is lower than 70 points, CLCVP technique will be initiated to improve the surgical conditions. At T5, the surgeon will re-evaluate the surgical field to assess the effectiveness of the CLCVP technique. At the same time, the surgeon will independently evaluate the performance of the anesthesiologist in controlling surgical field and ensuring the patient's safety, so as to comprehensively reflect the contribution of anesthesia management to the surgery. To ensure the objectivity of the assessment, the lead surgeon will remain blind to the patient group situation throughout the process.

   Secondary outcomes:
   * Cumulative consumption of nitroglycerine: Based on the criterion of CLCVP, record whether the patient needs to use nitroglycerine during the operation and the dose used.
   * Hemodynamic parameters: Collect data such as SBP, DBP, MAP, CVP, CO, SV, SVV, SVR, HR, SpO2 at the time when the patient enters the operating room (T0), after induction (T1), 15 minutes after adjusting the body position (T2), 30 minutes after the start of liver resection (T3), 60 minutes after the start of liver resection (T4), after liver resection (T5), and at the end of the operation (T6) to assess the influence of sildenafil on the intraoperative hemodynamic stability.
2. Safety evaluation indicators:

   * Blood gas analysis: Measure Hb, PH, and Lac at T1, T3, T4, and T5 to understand the patient's internal environment status.
   * Coagulation function：Understand the changes in the coagulation function of the patient during the operation by measuring the TEG of the patient at T2 and T5, and measure the APTT and PT values at D1, D3, and D5 to understand whether there is an impact on the patient's postoperative coagulation function after taking Sildenafil.
   * Intraoperative urine output: By recording the intraoperative urine output value of the patient at T6.
   * Adverse events in the recovery room：It is evaluated by measuring whether the patient has hypotension and whether there is hypoxemia in the recovery room.
   * Biochemical markers (Liver and kidney functions): It is evaluated by measuring the levels of TBil, Alb, AST, ALT, Cr, BUN of the patients on days -D1, D1, D3, and D5.
   * Complete blood count: At -D1, D1, D3, and D5, it is evaluated by measuring the patient's postoperative Hb, Plt, and Hct.
   * Cardiac function: By comparing the levels of BNP, CK-MB, and cTn of the patients on days D1 to assess whether Sildenafil has an impact on the patient's cardiac function.
   * Postoperative hospital stay and drainage indwelling time: Record the patient's hospital stay and drainage tube placement time to assess the patient's recovery speed.
   * Postoperative complications: Whether to enter the ICU after surgery, liver failure, bleeding, bile leakage, ascites, pleural effusion, and incision site infection.

     * (- D1: The day before surgery; - T0: half an hour before surgery; T0: entering the operating room; T1: post induction; T2: 5 minutes after 30° head-up and foot-down position; T3: 30 minutes after the start of liver resection; T4: 60 minutes after the start of liver resection; T5: after liver resection; T6: at the end of the operation; D1: Postoperative day 1; D3: Postoperative day 3; D5: Postoperative day 5)

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hepatic resection
* age from 18-85 years
* Child-Pugh ≤B
* ASA II-III
* willing to join the trial.

Exclusion Criteria:

* Pregnancy or Lactation
* Known Allergy to any Medications used in the Study
* Hemoglobin (Hb) < 90 g/L
* Body Mass Index (BMI) > 35 kg/m2 or < 18 kg/m2
* Hypertension > 180 mmHg
* Renal Impairment (Creatinine, Cr 178 µmol/L)
* Severe Cardiovascular Diseases including Active Coronary Artery Disease, Severe Valve Stenosis and Hypertrophic Obstructive Cardiomyopathy, History of Stroke Within Six Months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | At the end of the operation
  To quantify the IBL by calculating the amount of blood in the suction bottle (actual blood loss amount - saline irrigation amount) and the weight of the gauze blood pad ((weight of the gauze block after blood absorption in g - weight of the gauze block before blood absorption in g) / 1.054 (average density of blood in g/ml)).
The classification of the surgical field | At the end of the operation
  At T3 and T4, the surgeon will rate and score the liver surgical field according to Table 2. If the score is lower than 70 points, CLCVP technique will be initiated to improve the surgical conditions. At T5, the surgeon will re-evaluate the surgical field to assess the effectiveness of the CLCVP technique. At the same time, the surgeon will independently evaluate the performance of the anesthesiologist in controlling surgical field and ensuring the patient's safety, so as to comprehensively reflect the contribution of anesthesia management to the surgery. To ensure the objectivity of the assessment, the lead surgeon will remain blind to the patient group situation throughout the process.(At 30 minutes after the start of liver resection(T3), 60 minutes after the start of liver resection(T4) and after liver resection(T5))

SECONDARY OUTCOMES:
Cumulative consumption of nitroglycerine | At the end of the operation
  Based on the criterion of CLCVP, record whether the patient needs to use nitroglycerine during the operation and the dose used.
Hemodynamic parameters | At the end of the operation
  Collect data such as SBP, DBP, MAP, CVP, CO, SV, SVV, SVR, HR, SpO2 at the time when the patient enters the operating room (T0), after induction (T1), 15 minutes after adjusting the body position (T2), 30 minutes after the start of liver resection (T3), 60 minutes after the start of liver resection (T4), after liver resection (T5), and at the end of the operation (T6) to assess the influence of sildenafil on the intraoperative hemodynamic stability.
Blood gas analysis | At the end of the operation
  Measure Hb, PH, and Lac at T1, T3, T4, and T5 to understand the patient's internal environment status.(At post induction(T1), 5 minutes after 30° head-up and foot-down position(T2), 30 minutes after the start of liver resection(T3), 60 minutes after the start of liver resection(T4) and after liver resection(T5))
Intraoperative urine output | At the end of the operation(T6)
  By recording the intraoperative urine output value of the patient at T6.
Adverse events in the recovery room | After the end of surgery, Patient in recovery room.
  It is evaluated by measuring whether the patient has hypotension and whether there is hypoxemia in the recovery room.
Liver function | At the day before surgery(-D1), postoperative day 1(D1), postoperative day 3(D3) and postoperative day 5(D5).
  It is evaluated by measuring the levels of TBil, Alb, AST, ALT of the patients on days -D1, D1, D3, and D5.
kidney function | At the day before surgery(-D1), postoperative day 1(D1), postoperative day 3(D3) and postoperative day 5(D5).
  It is evaluated by measuring the levels of Cr, BUN of the patients on days -D1, D1, D3, and D5.
Complete blood count | At the day before surgery(-D1), postoperative day 1(D1), postoperative day 3(D3) and postoperative day 5(D5).
  At -D1, D1, D3, and D5, it is evaluated by measuring the patient's postoperative Hb, Plt, and Hct.
Cardiac function | At Postoperative day 1
  By comparing the levels of BNP, CK-MB, and cTn of the patients on days D1 to assess whether Sildenafil has an impact on the patient's cardiac function.
Postoperative hospital stay | At Postoperative day 5
  Record the patient's hospital stay to assess the patient's recovery speed.
Drainage indwelling time | At Postoperative day 5
  Record the drainage tube placement time to assess the patient's recovery speed.
Postoperative complications | At postoperative day 1, postoperative day 3 and postoperative day 5
  Whether to enter the ICU after surgery, liver failure, bleeding, bile leakage, ascites, pleural effusion, and incision site infection.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-ming Z Zhang, Principal Investigator — Chenzhou NO. 1 people's Hospital
Locations (1):
- Zhiming Zhang, Chenzhou, Hunan, China

REFERENCES:
- [Derived] Chen Q, Peng S, Zhou Y, Li S, Xu F, Yu Y, Wang P, Peng X, Zhao C, Xie A, Zhang Z. Perioperative sildenafil citrate administration in hepatectomy: a study protocol of randomized controlled trial. Trials. 2025 Jun 1;26(1):183. doi: 10.1186/s13063-025-08870-2. PMID 40450350